CLINICAL TRIAL: NCT03184662
Title: Randomized Trial to Assess the Efficacy of a High-intensity Physical Activity Program on Renal Function Decline in High Risk Patients With Type 2 Diabetes
Brief Title: Efficacy of a High-intensity Physical Activity Program on Renal Function in High Risk Patients With Type 2 Diabetes
Acronym: ACTIDIANE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID period
Sponsor: Poitiers University Hospital (Other)
Collaborators: University Hospital, Bordeaux (Other); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier Universitaire Dijon (Other); Centre Hospitalier Universitaire de Besancon (Other); Hopital Lariboisière (Other); Bichat Hospital (Other); Centre Hospitalier Sud Francilien (Other); University Hospital, Lille (Other); Centre Hospitalier Universitaire de Nice (Other); University Hospital, Caen (Other); University Hospital, Toulouse (Other); University Hospital, Tours (Other); Nantes University Hospital (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Hospices Civils de Lyon (Other); University Hospital, Montpellier (Other); University Hospital, Strasbourg (Other); Central Hospital, Nancy, France (Other); HOSPITAL, CHARTRES (Unknown); University of Liege (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTIDIANE
Record Dates: First submitted 2017-04-26; First posted 2017-06-12 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Type2 Diabetes; Diabetic Kidney Disease
Keywords: High-intensity physical activity; Diabetes; Renal function decline
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIPA group (Experimental): Twice weekly physical activity session in a dedicated structure, supervised by a graduated coach, alternating sessions of strengthening and intermittent HIPA, allowing a mixed stimulation of neuro-muscular and cardiovascular systems, and regular (every 3 months) adjustment of the intensity of the program.
  The sessions will be preferably performed in sports gyms but if required can also be performed online with supervised coaches, trained for the study.
  Interventions: Other: HIPA
- Control group (Active Comparator): Counseling of physical activity according to recommendations from the working group on Physical Activity of the SFD (French Language Diabetes Society).
  Interventions: Other: Counseling PA

INTERVENTIONS:
Other: HIPA — inclusion in a program with 2 weekly sessions of structured physical activity of 1 hour in a dedicated structure, under the supervision of a graduated coach.
  First 3 months : physical reconditioning 3 months and after: alternating sessions of physical strengthening and intermittent high-intensity physical activity Adaptation of the intensity of the program according to evaluation tests every 3 months
  Arms: HIPA group
Other: Counseling PA — Counseling of physical activity according to recommendations from the working group on Physical Activity of the SFD
  Arms: Control group

SUMMARY:
Type 2 diabetes is a chronic condition whose prevalence is increasing globally. Kidney disease is a key complication of diabetes and is among the most common cause of end-stage renal disease, requiring renal replacement therapy.

It has been shown that the trajectory of renal function (estimated glomerular filtration rate - eGFR) is of great prognostic value for renal and cardiovascular endpoints in diabetic patients. However the clinical use of this prognostic marker is not associated to date with a clear therapeutic intervention, effective in patients with type 2 diabetes identified with this biomarker.

In France, type 2 diabetes patients have twice less physical activity than non-diabetic persons. Recently, it has been published that physical activity was associated with an improvement of renal risk in patients with type 2 diabetes, recruited from the LOOK-AHEAD study. It was demonstrated that high-intensity physical activity (HIPA) can have several additional advantages over moderate-intensity, on blood pressure improvement, and cardiovascular risk profile modification. In addition, this procedure was shown to be safe in patients with high cardiovascular risk.

We plan to perform a randomized intervention comparing a structured program of high-intensity physical activity (HIPA) vs standard recommendations for physical activity on renal function decline (primary outcome) and mortality, renal and cardiovascular endpoints, patients' safety and quality of life (secondary outcomes). Study participants will be patients with established type 2 diabetes and a high renal risk, identified by rapid renal function decline, defined as a eGFR slope below -5ml/min per 1.73 m2/yr. The intervention is planned to last for 2 years.

DETAILED DESCRIPTION:
I- Visit organisation

V1 (screening) informed consent / examination / inclusion and non-inclusion criteria / medical history M/F LUTS / EPICES score / ECG Serum creatinine determination

V2 (Randomization) examination / verification of participation criteria / randomization Cystatin C collection / Biology Hypoglycemia notification / QAPPA / RPAQ / NAQA / Questionnaires (EQ-5D3L, SF12, Rosenberg Self esteem) / Accelerometer (ancillary) / Impedance-meter (ancillary) 6-minute step test / 10-meter walk test

V3 (1 month) examination / Hypoglycemia notification / QAPPA / RPAQ / Accelerometer (ancillary)

V4 (3 months) examination / Hypoglycemia notification / QAPPA / RPAQ / Questionnaires (EQ-5D3L, SF12, Rosenberg Self esteem) / Accelerometer (ancillary) 6-minute step test Biology

V5 (6 months) examination / Hypoglycemia notification / QAPPA / RPAQ / Questionnaires(EQ-5D3L, SF12, Rosenberg Self esteem) / Accelerometer (ancillary) 6-minute step test Cystatin C collection / Biology

V6 (12 months) examination / Hypoglycemia notification / QAPPA / RPAQ / NAQA / M/F LUTS / Questionnaires(EQ-5D3L, SF12, Rosenberg Self esteem) / ECG /Accelerometer (ancillary) / Impedance-meter (ancillary) Cystatin C collection / Biology 6-minute step test / 10-meter walk test

V7 (18 months) examination / Hypoglycemia notification / QAPPA / RPAQ / Questionnaires(EQ-5D3L, SF12, Rosenberg Self esteem) / Accelerometer (ancillary) Cystatin C collection / Biology 6-minute step test

V8 (24 months) / premature discontinuation examination / Hypoglycemia notification / QAPPA / RPAQ / NAQA / M/F LUTS / Questionnaires (EQ-5D3L, SF12, Rosenberg Self esteem) / ECG / Accelerometer (ancillary) / Impedance-meter (ancillary) 6-minute step test / 10-meter walk test Cystatin C collection / Biology

II- Recruitment criteria Inclusion

* Age : 45 and higher
* Female or male
* Type 2 diabetes with diabetes typing according to widely-accepted clinical and biological criteria [3].
* Subject able to practice physical activity. This includes a normal exercise test with or without anti-ischemic drugs, performed in the preceding 6 months or short before randomization. A certificate of no contre-indication for PA is to be delivered prior to randomization.
* With at least 3 available creatinine measurements in the 6 to 24 preceding months showing a rapid renal function decline defined as an eGFR slope below -5 ml/min/yr
* Estimated GFR equal to or higher than 30 ml/min/1.73m², defined by the CKD-EPI formula, at inclusion visit

Non inclusion

* Age strictly lower than 45 years
* Indication for cardiovascular rehabilitation (notably patient with ischemic heart disease or coronary revascularisation)
* Treatment with systemic NSAIDs or corticosteroids
* Lower limb amputation (above trans-metacarpal)
* Active proliferative retinopathy (risk of bleeding in case of effort)
* Contra-indication for the participation to PA:

  * Severe non-operated valvulopathy
  * Uncontrolled hypertension > 180/110 mmHg
  * Thrombus in the left ventricular cavity
  * Unstable coronaropathy, according to physician
  * NYHA stage IV heart failure
* Any condition that would jeopardize patient's safety or would affect the conduct of the study
* Pregnant or breast-feeding women or women of child-bearing potential without effective contraception during the study
* Any situation associated with unreliable cystatin-C determinations, according to patient medical history: HIV positivity, melanoma and thyroid dysfunction
* Simultaneous participation to any interventional study able to interfere with the current study endpoints
* Patients not registered to the social security
* Protected adults (under guardianship and trusteeship)
* Subject unable to express their consent (due to intellectual/mental incapacity)

III- Intervention HIPA group Twice weekly physical activity session in a dedicated structure, supervised by a graduated coach, alternating sessions of strengthening and intermittent HIPA, allowing a mixed stimulation of neuro-muscular and cardiovascular systems, and regular (every 3 months) adjustment of the intensity of the program.

Control group Counseling of physical activity according to recommendations from the working group on Physical Activity of the SFD (French Language Diabetes Society) supported by patient's oriented leaflet.

IV- Handling with the COVID-19 pandemics

The COVID-19 pandemics has modified the shape of the study with

* difficulties to comply with the study plan, including recruitment pace. Visits can be postponed if required but investigators are encouraged to follow the initial plan. The time between randomization and V3 (1 month) and V4 (3 months) can sometimes be too short and it is acceptable to perform this visit by phone or even to cancel it.
* difficulties to comply with physical activity (PA) plan. As PA facilities have been locked down in the pandemics context, the sports committee of the ACTIDIANE study has agreed to move attendances to the gym to some remote PA sessions, via websession or if not possible, via telephone coaching sessions.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Rapid renal decline function (yearly loss of eGFR over -5ml/min/1.73 m2) in the 6 to 24 preceding months

Exclusion Criteria:

* Lower limb amputation
* Indication for rehabilitation program
* Contra-indication for physical activity
* Unstable angina, left atrial thrombus,
* Unstable thyroid function
* Corticosteroids treatment
* Long-term NSAIDs
* Simultaneous participation to any interventional study able to interfere with the current study endpoints

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Renal Function Decline | 2 years
  Estimated glomerular filtration rate slope computed within 2 years, evaluated with the cystatin-derived CKD-EPI formula At least 3 available determinations of estimated glomerular filtration rate will be required to perform the calculation of the slope

SECONDARY OUTCOMES:
Incidence of ESRF | 2 years
  Incidence of end-stage renal failure requiring renal replacement therapy
Number of patients with a decrease in eGRF | 2 years
  Number of patients with a decrease in eGRF greater than 40% of baseline value
All cause death | 2 years
  Number of patients who died during the study (all cause)
Cardiovascular death | 2 years
  Cardiovascular death as proposed by the ICD-10 classification
Renal death | 2 years
  Renal death as defined as a situation where renal replacement therapy could be used but was not applied
MACE | 2 years
  MACE : major adverse cardiovascular endpoints : first occuring among cardiovascular death, myocardial infarction and stroke
Severe congestive heart failure | 2 years
  Severe congestive heart failure requiring hospitalization, adjudicated by a study outcome committee
Coronary artery disease | 2 years
  Coronary artery disease : myocardial infarction and/or coronary artery revascularizaton
Quality of life EQ-5D3L | 2 years
  Quality of life : assessed by using EQ-5D3L questionnaire
Male/Female lower urinary tract symptoms (LUTS) | 2 years
  Male/Female lower urinary tract symptoms : assessed by using M/F LUTS questionnaire
Safety of the intervention | 2 years
  including : adverse events, foot ulceration requiring medical advise, musculoskeletal disorders, hypoglycemia
Quality of life SF12 | 2 years
  Quality of life : assessed by using SF12 questionnaire
Safety of HIPA performed by e-coaching in the context of COVID infection | 2 years
  AE and SAE will be carefully reviewed to assess if the HIPA sessions are safe as performed with e-coaching/ telephone-coaching during lock-down due to the COVID-19 pandemics

CONTACTS AND LOCATIONS:
Locations (20):
- Hospital of Liège, Liège, Belgium
- France (19):
  - Besançon Hospital, Besançon
  - Bordeaux University Hospital, Bordeaux
  - Caen University Hospital, Caen
  - CH Chartres, Chartres
  - Clermont Ferrand University Hospital, Clermont-Ferrand
  - CHG Sud Francilien, Corbeil-Essonnes
  - CHU Dijon, Dijon
  - CHU Lille, Lille
  - Chu de Lyon, Lyon
  - CHRU, Montpellier
  - CHU Nancy, Nancy
  - Chu de Nice, Nice
  - Bichat University Hospital, Paris
  - La Riboisière Hospital, Paris
  - Hôpital Pitié Salpétrière, Paris
  - Poitiers University Hospital, Poitiers
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU de TOURS, Tours

IPD SHARING:
Plan to Share IPD: Yes
sharing policy is under the responsibility of the scientific committee who will organise this point Any request can be posted to the PI in the meantime.
Time Frame: pending
Access Criteria: pending
URL: https://actidiane.fr